CLINICAL TRIAL: NCT06950125
Title: Evaluation of the JUICE HA® as an Anti-sarcopenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CMUH114-REC3-004
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Sarcopenia in Elderly
Keywords: sarcopenia; quality of life
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: 60 participants aged 65 and above who have been diagnosed with sarcopenia will be randomly assigned into two groups using an envelope-drawing method: one group will receive the JUICE HA® supplement, while the other group will receive a placebo. The supplementation period will last for 12 weeks. Comparisons between the two groups will be conducted at baseline (pre-test) and after the intervention (post-test).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JUICE HA® supplement (Experimental): Bottle with 15 ml of JUICE HA® supplement
  Interventions: Other: JUICE HA® supplement
- Placebo (Placebo Comparator): Bottle of 15 mL liquid (non-effective product).
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Bottle of 15 mL liquid (non-effective product) will be taken once a day for 12 weeks.
  Arms: Placebo
Other: JUICE HA® supplement — Bottle of 15 mL JUICE HA® supplement will be taken once a day for 12 weeks.
  Arms: JUICE HA® supplement

SUMMARY:
This study plans to recruit 60 participants aged 65 years and older who have been diagnosed with sarcopenia by a physician. Participants will be randomly assigned into JUICE HA® supplement and placebo group. All of the participants will be asked to take 15 mL/day of JUICE HA® supplement or placebo group for 12 weeks. The aim of this trial is to evaluate the potential of JUICE HA® to enhance physiological status (muscle mass and functional fitness) and to improve the quality of life in patients with sarcopenia.

DETAILED DESCRIPTION:
JUICE HA® is a nutritional supplement formulated with hyaluronic acid (HA), branched-chain amino acids (BCAA), and chondroitin. Hyaluronic acid contributes to enhancing hydration levels in the skin and connective tissues; BCAA promotes muscle protein synthesis and repair; and chondroitin is believed to support the structural integrity and functionality of joints. The synergistic combination of these components is anticipated to provide comprehensive, multidimensional support for individuals with sarcopenia, potentially alleviating symptoms and improving overall quality of life. Therefore, this study will explore 15 mL/day of JUICE HA® supplement to improve the muscle mass and functional fitness in the elderly with sarcopenia.

This study aims to recruit 60 participants aged 65 years and older who have been diagnosed with sarcopenia by a physician and meet the Asian Working Group for Sarcopenia (AWGS) 2019 diagnostic criteria. Participants will be enrolled in a randomized control-group pretest-posttest design and randomly assigned to receive either the JUICE HA® supplement or a placebo (Lin et al., 2021). Functional fitness assessments, the Sarcopenia Quality of Life questionnaire (SarQoL), and blood sample collections will be conducted at baseline, at the 6th and 12th weeks of the supplementation period, and at the 6th and 12th weeks of the follow-up period. Blood samples will be analyzed for oxidative stress markers (SOD, MDA), inflammatory markers (TNF-α, IL-10), and muscle synthesis and degradation indicators (mTOR, MuRF1, atrogin-1). Body composition assessments will be performed at baseline, at the 12th week of the supplementation period, and at the 12th week of the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Participants that have been diagnosed with sarcopenia by a physician and meet the AWGS 2019 criteria for sarcopenia.

Exclusion Criteria:

* Participants with a history of severe lower extremity musculoskeletal injuries within the past six months or those who have a fear of blood sampling will be excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-13 (Estimated)

PRIMARY OUTCOMES:
Grip Strength | From enrollment to the end of treatment at 24 weeks
  Participants will be instructed to stand naturally with both arms relaxed at their sides. The examiner will adjust the grip span of the dynamometer, ensuring that when holding the handle, the second joint of the index finger forms approximately a 90-degree angle. Handgrip strength will be measured for both the dominant and non-dominant hands. After completing the measurement for one hand, the dynamometer will be reset to zero, and the participant will rest for 30 seconds before testing the other hand. Each hand will be tested twice, and the highest value recorded (in kilograms) will be used for analysis. Standard for male participants: < 28 kg; for female participants: < 18 kg.
Chair Stand Test | From enrollment to the end of treatment at 24 weeks
  Prior to data collection, participants will perform three practice trials to familiarize themselves with the test procedure. At the start of the test, participants will be seated on a chair with a neutral spine posture and both feet flat on the floor. Participants will be instructed to rise from the chair and return to a seated position as quickly as possible. The verbal cue "1, 2, 3, GO" will be given, and the stopwatch will be started simultaneously with the "GO" command. Participants will be instructed to complete five full sit-to-stand cycles as quickly as possible without using their arms for assistance. A total time exceeding 15 seconds is considered indicative of low muscle strength.
Appendicular Skeletal Muscle Mass (ASM) | From enrollment to the end of treatment at 24 weeks
  Appendicular skeletal muscle mass (ASM) will be measured using a Dual-Energy X-ray Absorptiometry (DXA) scanner. The skeletal muscle mass of the four limbs will be assessed to determine the participants' muscle status. A cut-off value of 20 kilograms for males and 15 kilograms for females will be used to define low muscle mass, with values below these thresholds indicating reduced skeletal muscle mass.
Appendicular Skeletal Muscle Mass Index | From enrollment to the end of treatment at 24 weeks
  The appendicular skeletal muscle mass (ASM) obtained from the DXA measurement will be divided by the square of the participant's height to calculate the appendicular skeletal muscle mass index (ASMI). A cut-off value of 7.0 kg/m² for males and 5.5 kg/m² for females will be used to define low muscle mass index, with values below these thresholds indicating low skeletal muscle mass relative to body size.
Gait Speed | From enrollment to the end of treatment at 24 weeks
  A 6-meter gait speed test will be conducted to assess walking speed. Participants will be instructed to walk at their usual pace over a distance of 6 meters, and the time taken to complete the distance will be recorded. Gait speed will be calculated by dividing the distance by the time, and a gait speed of less than 1.0 meter per second will be considered indicative of low physical performance.
Short Physical Performance Battery (SPPB) | From enrollment to the end of treatment at 24 weeks
  Researchers received training in the administration of the Short Physical Performance Battery (SPPB) and were audited by the same trainer to ensure accurate and standardized execution. The SPPB, with a total score of 12 points, comprises three components: a standing balance test, a gait speed test, and a chair stand test. Based on the total score, participants are classified as frail (4-7 points), pre-frail (8-9 points), or functionally normal (10-12 points). Before testing, researchers explained the procedures and purpose of the assessments to the participants and demonstrated the key points of each movement. Participants were allowed one practice trial before formal testing. A 3-minute rest period was provided between the practice and formal test for each component.
Sarcopenia Quality of Life (SarQoL) | From enrollment to the end of treatment at 24 weeks
  The Sarcopenia and Quality of Life (SarQoL) questionnaire will be used to assess the quality of life in individuals with sarcopenia. The questionnaire can be either self-administered by the participants or administered with the assistance of researchers through verbal questioning. The SarQoL consists of 55 items grouped into 22 questions and is designed to be completed within approximately 10 minutes.
Clinical Biochemistry of total antioxidant capacity and lipid peroxidation | From enrollment to the end of treatment at 24 weeks
  Blood samples were collected at five different time points (week 0, week 6, week 12, week 18, week 24). The scavenging ability of antioxidants (6-hydroxy-2,5,7,8-tetramethylchroman-2-carboxylic acid, Trolox) was determined using a curve, and the amount of Trolox equivalent to the test serum's inhibition rate was calculated. Next, the level of malondialdehyde (MDA), a standard biomarker of lipid peroxidation, was determined by an ELISA kit provided by the Caman Company (Cayman Chemical Company, Michigan, USA). As described in the protocol, the reaction mixture was boiled at 90-100°C for 60 min, and the absorbance at 550 nm was measured using an ELISA plate reader (Tecan GENios, A-5082, Austria). The values are expressed as micromoles of MDA per liter.
Clinical Biochemistry of the inflammatory response | From enrollment to the end of treatment at 24 weeks
  Blood samples were collected at five different time points (week 0, week 6, week 12, week 18, week 24). The concentrations of serum cytokines IL-6, IL-10, TNF-α, and high-sensitivity C-reactive protein (hs-CRP) will be measured using commercially available assay kits (Bio-Legend Inc., No. 430207, San Diego, CA) and enzyme-linked immunosorbent assay (ELISA) methods (Tecan GENios, A-5082, Austria). Absorbance readings will be taken at wavelengths of 450 nm, 545 nm, 520 nm, and 570 nm, respectively. The concentrations of IL-6, IL-10, TNF-α, and hs-CRP in serum samples will be calculated based on the corresponding standard curves.
Clinical Biochemistry of biomarkers of muscle synthesis and degradation | From enrollment to the end of treatment at 24 weeks
  Blood samples were collected at five different time points (week 0, week 6, week 12, week 18, week 24). Then will be assessed by measuring serum levels of mTOR and RSK (muscle synthesis markers) and MuRF1 and atrogin-1 (muscle degradation markers). These biomarkers will be quantified using commercially available assay kits and enzyme-linked immunosorbent assay (ELISA) methods (Tecan GENios, A-5082, Austria). Absorbance readings will be taken at wavelengths of 450 nm and 570 nm, respectively. The concentrations of mTOR, RSK, MuRF1, and atrogin-1 in serum samples will be determined based on the corresponding standard curves.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No